CLINICAL TRIAL: NCT00735592
Title: The Study Intend to Evaluate the Usefulness of Performing a Follow up X Rays in Children Admitted With Lobar Pneumonia.
Brief Title: Value of Radiological Follow up in Children Hospitalized With Lobar Pneumonia
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0012-08-EMC
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Pneumonia
Keywords: X rays findings
MeSH Terms: conditions — Pneumonia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Children discharged with the recommendation of performing a follow up X rays after lobar pneumonia
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Retrospective data obtained from electronic files

SUMMARY:
The study intends to assess the utility of performing a follow up X rays in children admitted to pediatric wards with lobar pneumonia. Usually those children are discharged with a recommendation for a follow up X rays but there are no enough studies proving that this recommendation is really necessary.

DETAILED DESCRIPTION:
Thew study will include follow up data in a group of about 200 patients admitted with lobar pneumonia during the years 2006 to 2007. All the clinical and laboratory data will be collected and also the X rays findings.

The findings of follow up X rays if they were performed will also be summarized.

ELIGIBILITY:
Inclusion Criteria: All pediatric patients discharged with the diagnosis of lobar pneumonia.

Exclusion Criteria: Patients with diagnosis of chronic diseases.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients admitted during the years 2006 and 2007 with the diagnosis of lobar pneumonia.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sakran Waheeb, MD, Principal Investigator — Pediatric Dpt B - Ha'Emek Medical Center - Afula - 18101 - Israel; Ronza Andraws, MD, Principal Investigator — Pediatric Dpt B - Ha'Emek Medical Center - Afula - Israel
Locations (1):
- Pediatric Dpt B - Ha'Emek Medical Center, Afula, Afula, Israel